CLINICAL TRIAL: NCT05681455
Title: Physiotherapy for Persistent Function by Superficial Neuromodulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Physiotherapy for Persistent Function by Superficial Neuromodulation, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22/32
Record Dates: First submitted 2022-12-05; First posted 2023-01-12 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Post-Acute COVID-19 Syndrome; Dysautonomia; Neuromodulation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Autonomic Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: triple-blind randomized controlled clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A two-phase microcurrent with a frequency between 1.14 Hertz and 14.29 Hertz and currents between 0.1 and 0.9 mA will be applied.
  A total of 15 sessions in 7.5 weeks. Twice a week. The session time with microcurrents will last 60 minutes.
  Interventions: Device: Neuromodulation NESA NXSIGNAL® device
- Placebo group (Placebo Comparator): Microcurrent machines shall be operated in such a way that they have a light signal but do not emit current. Neither the physical therapists who place them nor the subjects will be able to distinguish current-emitting machines from placebo machines.
  A total of 15 sessions in 7.5 weeks. Twice a week. The session time with placebo will last 60 minutes.
  Interventions: Device: Neuromodulation NESA NXSIGNAL® device

INTERVENTIONS:
Device: Neuromodulation NESA NXSIGNAL® device — Good positioning of the NXSIGNAL® device, as well as proper programming, is of vital importance for the achievement of the objective. General guidelines will be established, which should always be followed with the application of NESA microcurrents, and specific guidelines for this particular study, in order to obtain as homogeneous a sample as possible and to bring the device programming as close as possible to the objective to be pursued in the clinical trial. General guidelines for the application of XSIGNAL®.
  The skin should be clean, free of creams and grease, so it will be necessary to clean with alcohol or similar. The placement of the gloves and socks of the device should follow the established protocols, paying attention to the location of each semielectrode in its anatomical position. The device has a color system to determine the location of each wire.
  The directional electrode will be placed in the cervical area at the superficial level between C6 and C7.

SUMMARY:
Objectives:

To evaluate pressure pain thresholds, fatigue scales, quality of life and sleep quality, in women with Persistent Covid (PC), pre- and post-treatment using electrotherapy and in a placebo group of PC patients.

Relevance:

This trial can be a tool for patients affected by CP who present pain and fatigue problems, insomnia or signs of imbalance of their Autonomic Nervous System. It aims to improve their rest and recovery for a better quality of life that allows them to recover their Activities of Daily Living.

We have designed the study with a commitment to placebo group treatment after completion, if positive results are obtained.

A 6-month and 1-year follow-up will be scheduled.

Secondary objectives:

To analyze the effects on quality of life, fatigue and sleep. To analyze the presence of cardiac variability and pre- and post-treatment cortisol values.

Patients and Methods:

12 patients with CP will receive 15 sessions of electrotherapy. 12 will receive a placebo.

Mechanical sensitivity pre-post, by means of an algometer, cardiac variability, cortisol levels, and other variables, will be measured by means of questionnaires.

Mechanical sensitivity to pain will be measured using an algometer (Baseline 12-0300 MMT). Patients will be instructed to report when the sensation of pressure changes to pain.

The pre-post electrotherapy treatment described above will be measured, the differences in mechanical sensitivity, pain threshold to pressure, the Pittsburg questionnaires, SF-36, MFIS and EQooL-5.

Follow-up will be done at 6 months and at one year. The study design is a triple-blind randomized controlled clinical trial. Patients who sign the consent form will be evaluated by an internist who will perform a physical examination at the clinic of the Faculty of Nursing and Physiotherapy of the Pontifical University of Salamanca (UPSA).

The sample will be randomized. 12 patients will receive treatment and 12 patients will receive a placebo. With a commitment to treat these patients in the event that positive results are obtained after the end of the study.

A biphasic microcurrent will be applied with a frequency between 1.14 Hertz and 14.29 Hertz and intensities between 0.1 and 0.9 mA.

Frequency: 2 times a week. A total of 15 sessions in 7.5 weeks. The session time with microcurrents will last 60 minutes.

.

ELIGIBILITY:
Inclusion Criteria:

* Women who have had symptoms of PC for more than one year.
* Signs of central sensitization.

Exclusion Criteria:

* Previous treatment with surgery.
* Previous spinal trauma.
* Whiplash.
* Pregnancy situation.
* Previous musculoskeletal disease (rheumatoid arthritis, sympathetic-reflex dystrophy, fibromyalgia).
* Pacemaker.
* Electric drug pump.
* Skin sensitivity alterations.
* Analgesic or anxiolytic drug treatment during the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain Pressure Threshold | Change from Baseline Pain Pressure Threshold at 1 year
  Central sensitization by assessment of the Pressure Pain Threshold (PPU) in kg: Baseline 12-0300 MMT algometer at cervical C5-C6, dorsal D5-D6 and anterior tibial muscle.

SECONDARY OUTCOMES:
Quality of life RELATED TO HEALTH | Change from baseline quality of life related to health at 1 year
  SF-36 questionnaire
Quality of life RELATED TO HEALTH | Change from baseline quality of life related to health at 1 year
  EuroQool-5-D questionnaire
effects on fatigue | Change from Baseline fatigue at 1 year
  MFIS questionnaire (Modificated Fatigue Impact Scale)
Quality of sleep | Change from Baseline Quality of Sleep at 1 year
  Pittsburg questionnaire
cardiac variability | Change from Baseline Cardiac variability at 1 year
  HRV (cardiac variability)" in ms 2. "SDNN (Standard deviation of all R-R intervals)" in ms 3. "rMSSD (Root mean square of the union of adjacent R-R intervals)" in ms
Cortisol levels | Change from Baseline Cortisol level at 1 year
  Soma OFCII cube device in nmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy, Occupational Therapy, Rehabilitation and Physical Medicine. Faculty of Health Sciences. Rey Juan Carlos University, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaber TAK, Ashish A, Unsworth A. Persistent post-covid symptoms in healthcare workers. Occup Med (Lond). 2021 Jun 16;71(3):144-146. doi: 10.1093/occmed/kqab043. PMID 33830208
- [Result] Burgess LC, Venugopalan L, Badger J, Street T, Alon G, Jarvis JC, Wainwright TW, Everington T, Taylor P, Swain ID. Effect of neuromuscular electrical stimulation on the recovery of people with COVID-19 admitted to the intensive care unit: A narrative review. J Rehabil Med. 2021 Mar 18;53(3):jrm00164. doi: 10.2340/16501977-2805. PMID 33634830
- See also: Related Info — https://www.semg.es/index.php/consensos-guias-y-protocolos/363-guia-clinica-para-la-atencion-al-paciente-long-covid-covid-persistente